CLINICAL TRIAL: NCT00663052
Title: A Randomized, Double-Blind Trial Assessing the Efficacy and Safety of Etanercept 50 mg Twice Weekly and Etanercept 50 mg Once Weekly for the Treatment of Moderate to Severe Psoriasis
Brief Title: Study Evaluating Etanercept for the Treatment of Moderate to Severe Psoriasis
Acronym: PRISTINE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 0881A6-4425; B1801013
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Results first posted 2012-04-23 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-03

CONDITIONS: Plaque Psoriasis; Psoriasis
Keywords: Enbrel; Psoriasis; Topical Psoriasis; Wyeth Psoriasis; Active Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): A
  Interventions: Drug: Etanercept
- Group B (Experimental): B
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — ETN 50 mg QW + PBO QW for 12 weeks followed by ETN 50 mg QW for 12 weeks.
  Arms: Group A
Drug: Etanercept — ETN 50 mg BIW for 12 weeks folowed ETN 50 mg QW for 12 weeks.
  Arms: Group B

SUMMARY:
The purpose of this study is to compare the safety and efficacy of different doses of etanercept for the treatment of moderate to severe psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at time of consent.
* Active, moderate to severe chronic plaque psoriasis defined by the following criteria: Clinically stable, plaque psoriasis involving greater than or equal to 10% body surface area (BSA) or PASI greater than or equal to 10.
* In the opinion of the investigator, failure, intolerance, contraindication or not a candidate for the following: Methotrexate (MTX), cyclosporine and psoralen plus ultraviolet A radiation (PUVA) therapy.

Exclusion Criteria:

* Evidence of skin conditions (e.g., eczema) other than psoriasis that would interfere with evaluations of the effect of study medication on psoriasis.
* Rheumatologic disease such as rheumatoid arthritis, systemic lupus erythematous, systemic vasculitis, scleroderma and polymyositis, or associated syndromes.
* Active or recent (within 2 years) tuberculosis (TB) infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2008-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (36):
- Argentina (2):
  - Pfizer Investigational Site, Capital Federal, Buenos Aires
  - Pfizer Investigational Site, San Miguel, Buenos Aires
- Austria (2):
  - Pfizer Investigational Site, Feldkirch
  - Pfizer Investigational Site, Vienna
- Belgium (3):
  - Pfizer Investigational Site, Brussels, Belgium
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Liège
- Czechia (3):
  - Pfizer Investigational Site, Jihlava
  - Pfizer Investigational Site, Ostrava- Poruba
  - Pfizer Investigational Site, Plzen-Bory
- Germany (7):
  - Pfizer Investigational Site, Bochum
  - Pfizer Investigational Site, Erlangen
  - Pfizer Investigational Site, Frankfurt am Main
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Kiel
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Osnabrück
- Pfizer Investigational Site, Athens, Greece
- Hungary (4):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Debrecen
  - Pfizer Investigational Site, Miskolc
  - Pfizer Investigational Site, Szeged
- Italy (2):
  - Pfizer Investigational Site, Catanzaro
  - Pfizer Investigational Site, L’Aquila
- Mexico (3):
  - Pfizer Investigational Site, Zapopan, Jalisco
  - Pfizer Investigational Site, Monterrey, Nuevo Leon / Mexico
  - Pfizer Investigational Site, Monterrey, Nuevo León
- South Korea (2):
  - Pfizer Investigational Site, Gangnam-gu
  - Pfizer Investigational Site, Seoul
- Spain (4):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Santiago de Compostela, La Coruña
  - Pfizer Investigational Site, Fuenlabrada, Madrid
  - Pfizer Investigational Site, Valencia
- Taiwan (2):
  - Pfizer Investigational Site, Taipei
  - Pfizer Investigational Site, Taipei TOC
- Pfizer Investigational Site, Bangkok, Thailand

REFERENCES:
- [Derived] Kemeny L, Amaya M, Cetkovska P, Rajatanavin N, Lee WR, Szumski A, Marshall L, Mahgoub EY, Aldinc E. Effect of etanercept therapy on psoriasis symptoms in patients from Latin America, Central Europe, and Asia: a subset analysis of the PRISTINE trial. BMC Dermatol. 2015 May 21;15:9. doi: 10.1186/s12895-015-0028-8. PMID 25994179
- [Derived] Griffiths CE, Christophers E, Szumski A, Jones H, Mallbris L. Impact of early vs. late disease onset on treatment response to etanercept in patients with psoriasis. Br J Dermatol. 2015 Nov;173(5):1271-3. doi: 10.1111/bjd.13865. Epub 2015 Aug 17. No abstract available. PMID 25913550
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881A6-4425&StudyName=Study%20Evaluating%20Etanercept%20for%20the%20Treatment%20of%20Moderate%20to%20Severe%20Psoriasis

RESULTS

PARTICIPANT FLOW:
Groups:
- ETN 50 mg BW/QW: Etanercept (ETN) subcutaneously (s.c.) 50 milligram (mg) twice weekly (BIW) for 12 weeks (double blind phase) followed by ETN s.c. 50 mg once weekly (QW) for 12 weeks (open label Phase).
- ETN 50 mg QW/QW: ETN s.c. 50 mg QW and matching placebo for ETN QW for 12 weeks (double blind phase), followed by ETN s.c. 50 mg QW for 12 weeks (open label phase).
Period: Overall Study
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Started | 136 | 137
Completed | 124 | 127
Not Completed | 12 | 10
Not completed — Adverse Event | 6 | 3
Not completed — Discontinuation of Study by Sponsor | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Unsatisfactory Response - Efficacy | 1 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW | Total
Number analyzed (Participants) | 136 | 137 | 273
Age Continuous [Mean (Standard Deviation); unit: Years] | 43.95 (12.68) | 43.85 (12.69) | 43.90 (12.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 36 | 83
  Male | 89 | 101 | 190
Mean Psoriasis Area and Severity Index (PASI) Score [Mean (Standard Deviation); unit: Units on scale] — PASI: Combined assessment of lesion severity and area affected into single score; range: 0(no disease) to 72(maximal disease). Body was divided into 4 sections (head, arms, trunk, legs); each area was scored by itself and scores were combined for final PASI.
  Units on scale | 21.4 (9.4) | 20.9 (9.4) | 21.2 (9.4)
Number of Participants Achieving the Physician Global Assessment (PGA) of Psoriasis Reponses [Number; unit: Participants] — PGA of Psoriasis: score based on dermatologist's assessment of head, scalp, and neck psoriasis (averaged over all lesions). The PGA of Psoriasis scale ranges from 0 (no psorasis) to 5 (severe disease). PGA score of 0 = Status of Clear; 1 = Almost Clear and 2 = Mild.
  Participants
    PGA Clear (0) | 0 | 0 | 0
    PGA Clear/Almost Clear (0,1) | 0 | 1 | 1
    PGA Clear/Almost Clear/Mild (0,1,2) | 13 | 17 | 30
Percent Body Surface Area (BSA) of Involvement [Mean (Standard Deviation); unit: Percentage of BSA] | 33.0 (19.4) | 32.9 (21.0) | 33.0 (20.2)
Number of Participants Not Using Topical Preparations [Number; unit: Participants] — Moderate topical steroids to very potent topical steroids, topical vitamin D analogs, topical steroids in combination with vitamin D analogs, and anthralin compounds were prohibited for 14 days before the baseline visit until week 12.
  Participants | 120 | 124 | 244
Number of Participants Evaluated Using Psoriasis Physician Satisfaction Questionnaire (PPSQ) [Number; unit: Participants] — PPSQ includes two global satisfaction questions to which physicians respond either 'satisfactory' or 'not satisfactory'.
  Participants
    Consider patient's condition satisfactory | 16 | 16 | 32
    Consider primary psoriasis therapy satisfactory | 15 | 17 | 32
Mean Psoriasis Subject Satisfaction Questionnaire (PSSQ) Scores [Mean (Standard Deviation); unit: Units on scale] — PSSQ: participant's assessment which includes 18 items, 16 items (1-16) scored using Likert score with scores from 0 (very dissatisfied) to 4 (very satisfied) and 5 (never had this problem). Only those participants who do not have score of 5 at baseline were included in the item 1-16 analyses. Two items (17, 18) are with Yes/No answers.
  Units on scale
    Overall appearance of your skin | 0.9 (0.8) | 0.9 (0.9) | 0.9 (0.9)
    Flaking skin | 1.0 (0.9) | 1.0 (0.9) | 1.0 (0.9)
    Skin redness | 1.1 (0.9) | 1.0 (0.9) | 1.0 (0.9)
    Skin tightness | 1.2 (0.9) | 1.2 (1.0) | 1.2 (1.0)
    Skin bleeding | 1.7 (1.0) | 1.8 (1.2) | 1.7 (1.1)
    Burning sensation in the skin | 1.5 (1.1) | 1.5 (1.1) | 1.5 (1.1)
    Skin pain | 1.5 (1.2) | 1.5 (1.1) | 1.5 (1.1)
    Joint pain | 1.8 (1.3) | 1.8 (1.4) | 1.8 (1.3)
    Comfort level with your appearance | 1.3 (1.1) | 1.2 (1.0) | 1.3 (1.0)
    Anxiety | 1.8 (1.1) | 1.7 (1.1) | 1.7 (1.1)
    Depression | 2.0 (1.1) | 1.9 (1.1) | 1.9 (1.1)
    Fatigue | 2.0 (1.0) | 1.8 (1.0) | 1.9 (1.0)
    How others respond to your appearance | 1.6 (1.0) | 1.8 (1.0) | 1.7 (1.0)
    How your skin affects social, leisure activities | 1.5 (1.2) | 1.3 (1.0) | 1.4 (1.1)
    Satisfaction with psoriasis treatment in general | 1.4 (1.2) | 1.4 (1.1) | 1.4 (1.1)
    Would like to continue with my current treatment | 2.0 (1.6) | 2.2 (1.6) | 2.1 (1.6)
Number of Participants Who were Considered Satisfied According to Psoriasis Subject Satisfaction [Number; unit: Participants] — PSSQ: participant's assessment which includes 18 items, 16 items (1-16) scored using Likert score with scores from 0 (very dissatisfied) to 4 (very satisfied) and 5 (never had this problem). Only those participants who do not have score of 5 at baseline were included in the item 1-16 analyses. Two items (17, 18) are with Yes/No answers.
  Participants
    Satisfaction with health state | 25 | 28 | 53
    Satisfaction with primary psoriasis treatment | 31 | 28 | 59
Mean Dermatology Life Quality Index (DLQI) Total Score [Mean (Standard Deviation); unit: Units on scale] — DLQI is the dermatology-specific quality of life measure used for psoriatic population. The 10-item questionnaire has a score range of 0 to 30 with higher scores indicating poor quality of life. An estimate of the minimal clinically important difference of the DLQI total score is a 5 point improvement. Total score range: 0 (best) to 30 (worst).
  Units on scale | 14.1 (7.3) | 15.0 (8.0) | 14.6 (7.7)
Mean Euro Quality of Life 5 Dimension (EQ-5D) Utility Index Scores [Mean (Standard Deviation); unit: Units on scale] — EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains; 1 indicates better health state (no problems); 3 indicates worst health state (example "confined to bed").
  Units on scale | 0.65 (0.30) | 0.66 (0.31) | 0.65 (0.31)
Mean Hospital Anxiety and Depression Scale (HADS) Anxiety and Depression Scores [Mean (Standard Deviation); unit: Units on scale] — HADS: participant rated questionnaire with 2 subscales for anxiety and depression. Each subscale comprised of 7 items with range 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). Total score 0 to 21 for each subscale; higher score indicates greater severity of anxiety and depression symptoms.
  Units on scale
    HADS Anxiety Score | 7.2 (4.4) | 6.9 (4.1) | 7.0 (4.3)
    HADS Depression Score | 6.0 (4.1) | 6.5 (4.1) | 6.2 (4.1)
Work Productivity and Activity Impairment: Psoriasis (WPAI:PSO) [Mean (Standard Deviation); unit: Percentage of indicated parameter] — WPAI:PSO - participant rated questionnaire to assess effect of psoriasis on ability to work and perform regular activities in 4 areas: percent activity impairment (0 [no effect on daily activities] to 100 [psoriasis completely prevented from doing daily activities]), percent impairment while working (0 [no effect] to 100 [completely prevented from working]); percent work time missed due to psoriasis, and percent overall work impairment (0 [no effect] to 100 [completely prevented from working]).
  Percentage of indicated parameter
    Percent Activity Impairment Due to Problem | 39.77 (28.96) | 40.15 (30.94) | 39.96 (29.93)
    Percent Impairment While Working Due to Problem | 24.36 (23.28) | 26.09 (27.08) | 25.27 (25.29)
    Percent Overall Work Impairment Due to Problem | 25.45 (23.53) | 29.51 (28.66) | 27.54 (26.30)
    Percent Work Time Missed | 3.60 (16.14) | 7.19 (18.92) | 5.45 (17.67)
Mean Medical Outcomes Study (MOS) Sleep Scale Scores [Mean (Standard Deviation); unit: Units on scale] — MOS scale has 12 questions to assess sleep quality & quantity: 1)time to fall asleep, 2)hours of sleep/night in past 4 weeks,3)sleep not peaceful, 4)got enough sleep to feel rested in morning,5)awaken short of breath/headache 6)feel drowsy in day,7)trouble going to sleep, 8)wake up during sleep; trouble going back to sleep,9)trouble staying awake in day, 10)Snoring,11)take naps in day,12)get amount of sleep needed. Sleep problem index(SPI) I:mean of 4,5,7,8,9,12; SPI II:mean of 1,3,4,5,6,7,8,9,12. All reported responses are on scale:0-100, higher scores indicate greater intensity of attribute.
  Units on scale
    Sleep Snoring | 37.9 (29.6) | 45.7 (31.0) | 41.9 (30.5)
    Sleep Somnolence | 29.9 (19.9) | 30.9 (19.3) | 30.4 (19.5)
    Sleep Short of Breath or Headache | 13.2 (20.4) | 14.3 (20.7) | 13.8 (20.5)
    Sleep Adequacy | 54.6 (25.9) | 54.0 (27.3) | 54.3 (26.6)
    Sleep Disturbance | 35.0 (23.6) | 34.4 (23.8) | 34.7 (23.6)
    Sleep Quantity | 6.9 (1.4) | 6.9 (1.4) | 6.9 (1.4)
    Sleep Problem Index I | 32.5 (18.7) | 32.9 (19.1) | 32.7 (18.9)
    Sleep Problem Index II | 33.9 (18.2) | 34.2 (19.6) | 34.0 (18.9)
Mean Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Questionnaire Total Scores [Mean (Standard Deviation); unit: Units on scale] — FACIT Fatigue questionnaire: Participant rated 13- item questionnaire to assess fatigue. For each question, participant rates his / her condition for the past week on a 5-point Likert scale ranging from 0 (not at all) to 4 (very much). Higher scores always represent less fatigue (Total score range= 0 to 52).
  Units on scale | 37.9 (10.0) | 36.7 (10.8) | 37.3 (10.4)
Number of Participants With Emergency Room Visits [Number; unit: Participants] | 6 | 8 | 14
Mean Number of Emergency Room Days [Mean (Standard Deviation); unit: Days] | 7.8 (5.64) | 9.4 (7.31) | 8.7 (6.45)
Number of Participants With Doctor Visits [Number; unit: Participants] | 58 | 61 | 119
Mean Number of Doctor Visits [Mean (Standard Deviation); unit: Visits] | 2.9 (3.36) | 3.0 (3.68) | 3.0 (3.51)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a 75% Improvement From Baseline in Psoriasis Area and Severity Index (PASI) Score at Week 24
Description: PASI: Combined assessment of lesion severity and area affected into single score; range: 0(no disease) to 72(maximal disease). Body was divided into 4 sections (head, arms, trunk, legs); each area was scored by itself and scores were combined for final PASI. For each section percent area of skin involved was estimated: 0 (0%) to 6 (90 - 100%), and severity was estimated by clinical signs: erythema, induration, and desquamation; scale: 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each section * area score * weight of section (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4).
Time Frame: Week 24
Population: Modified intent-to-treat (mITT) population: all randomly assigned participants who received at least 1 ETN dose and had both baseline and on-therapy PASI evaluations. If participant had a missing evaluation for any time point assessments, the last observation carried forward (LOCF) method of imputation was used.
Measure: Number; unit: Percentage of participants
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Percentage of participants | 78.2 | 59.9
Statistical Analysis 1: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; With 125 participants/group, estimation was: 1)approximately 90% power to reject null hypothesis- PASI 75 response rate at 24 weeks: 50% in ETN 50 mg QW, assuming true rate is 65% or greater; 2)90% power to reject null hypothesis- PASI 75 response rate at 24 weeks: 60% in 50 mg BIW, assuming true rate is 74% or greater. The 95% CI widths on these are approximately ±8.8%, indicating PASI 75 for ETN 50 mg QW and ETN 50 mg BIW must be at least 58.8% & 68.8%, respectively to reject null hypotheses; Test type: Superiority or Other; p = 0.0015, Fisher Exact; Proportion difference = 18.34, 95% CI 2-sided [6.80 to 29.88] — Primary endpoint used 95% CI to compare to prespecified target rates for each treatment arm

2. Secondary Outcome: Percentage of Participants Achieving a 50% Improvement From Baseline in Psoriasis Area and Severity Index (PASI) Score at Each Visit Through Week 24
Description: as for outcome 1
Time Frame: Baseline to Week 24
Population: mITT population: all randomly assigned participants who received at least 1 ETN dose and had both baseline and on-therapy PASI evaluations. If participant had a missing evaluation for any time point assessments, the LOCF method of imputation was used.
Measure: Number; unit: Percentage of participants
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Percentage of participants
  Week 2 | 9.0 | 5.9
  Week 4 | 38.3 | 20.4
  Week 8 | 71.4 | 51.8
  Week 12 | 88.0 | 67.9
  Week 16 | 92.5 | 78.1
  Week 20 | 93.2 | 82.5
  Week 24 | 92.5 | 81.0
Statistical Analysis 1: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 2; Test type: Superiority or Other; p = 0.3605, Fisher Exact; Proportion difference = 3.14, 95% CI 2-sided [-3.88 to 10.16]
Statistical Analysis 2: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 4; Test type: Superiority or Other; p = 0.0013, Fisher Exact; Proportion difference = 17.91, 95% CI 2-sided [6.50 to 29.32]
Statistical Analysis 3: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 8; Test type: Superiority or Other; p = 0.0011, Fisher Exact; Proportion difference = 19.60, 95% CI 2-sided [7.51 to 31.70]
Statistical Analysis 4: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 12; Test type: Superiority or Other; p < .0001, Fisher Exact; Proportion difference = 20.09, 95% CI 2-sided [9.77 to 30.40]
Statistical Analysis 5: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 16; Test type: Superiority or Other; p = 0.0010, Fisher Exact; Proportion difference = 14.38, 95% CI 2-sided [5.39 to 23.37]
Statistical Analysis 6: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 20; Test type: Superiority or Other; p = 0.0087, Fisher Exact; Proportion difference = 10.75, 95% CI 2-sided [2.35 to 19.16]
Statistical Analysis 7: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 24; Test type: Superiority or Other; p = 0.0068, Fisher Exact; Proportion difference = 11.46, 95% CI 2-sided [2.77 to 20.15]

3. Secondary Outcome: Percentage of Participants Achieving a 75% Improvement From Baseline in Psoriasis Area and Severity Index (PASI) Score at Each Visit Through Week 24
Description: as for outcome 1
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Percentage of participants
  Week 2 | 1.5 | 0.0
  Week 4 | 6.0 | 4.4
  Week 8 | 35.3 | 21.9
  Week 12 | 62.4 | 37.2
  Week 16 | 72.9 | 51.1
  Week 20 | 78.2 | 58.4
  Week 24 | 78.2 | 59.9
Statistical Analysis 1: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 2; Test type: Superiority or Other; p = 0.2435, Fisher Exact; Proportion difference = 1.50, 95% CI 2-sided [-1.31 to 4.32]
Statistical Analysis 2: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 4; Test type: Superiority or Other; p = 0.5929, Fisher Exact; Proportion difference = 1.64, 95% CI 2-sided [-4.40 to 7.67]
Statistical Analysis 3: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 8; Test type: Superiority or Other; p = 0.0156, Fisher Exact; Proportion difference = 13.44, 95% CI 2-sided [2.02 to 24.86]
Statistical Analysis 4: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 12; Test type: Superiority or Other; p < .0001, Fisher Exact; Proportion difference = 25.18, 95% CI 2-sided [12.89 to 37.47]
Statistical Analysis 5: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 16; Test type: Superiority or Other; p = 0.0003, Fisher Exact; Proportion difference = 21.84, 95% CI 2-sided [9.82 to 33.85]
Statistical Analysis 6: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 20; Test type: Superiority or Other; p = 0.0006, Fisher Exact; Proportion difference = 19.80, 95% CI 2-sided [8.23 to 31.38]
Statistical Analysis 7: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 24; Test type: Superiority or Other; p = 0.0015, Fisher Exact; Proportion difference = 18.34, 95% CI 2-sided [6.80 to 29.88]

4. Secondary Outcome: Percentage of Participants Achieving a 90% Improvement From Baseline in Psoriasis Area and Severity Index (PASI) Score at Each Visit Through Week 24
Description: as for outcome 1
Time Frame: Baseline to week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Percentage of participants
  Week 2 | 0.0 | 0.0
  Week 4 | 0.8 | 0.7
  Week 8 | 9.8 | 5.8
  Week 12 | 29.3 | 10.9
  Week 16 | 42.9 | 25.5
  Week 20 | 45.1 | 29.2
  Week 24 | 49.6 | 32.8
Statistical Analysis 1: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 2; Test type: Superiority or Other; Fisher Exact — The P-value at Week 2 was not applicable as the percentage of participants achieving 90% improvement in PASI in both treatment groups were 0%; Proportion difference = 0.00, 95% CI 2-sided [-0.74 to 0.74]
Statistical Analysis 2: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 4; Test type: Superiority or Other; p = 1.0000, Fisher Exact; Proportion difference = 0.02, 95% CI 2-sided [-2.77 to 2.81]
Statistical Analysis 3: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 8; Test type: Superiority or Other; p = 0.2611, Fisher Exact; Proportion difference = 3.94, 95% CI 2-sided [-3.20 to 11.07]
Statistical Analysis 4: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 12; Test type: Superiority or Other; p = 0.0002, Fisher Exact; Proportion difference = 18.37, 95% CI 2-sided [8.30 to 28.45]
Statistical Analysis 5: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 16; Test type: Superiority or Other; p = 0.0031, Fisher Exact; Proportion difference = 17.31, 95% CI 2-sided [5.43 to 29.19]
Statistical Analysis 6: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 20; Test type: Superiority or Other; p = 0.0081, Fisher Exact; Proportion difference = 15.92, 95% CI 2-sided [3.80 to 28.04]
Statistical Analysis 7: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 24; Test type: Superiority or Other; p = 0.0064, Fisher Exact; Proportion difference = 16.78, 95% CI 2-sided [4.46 to 29.10]

5. Secondary Outcome: Percentage of Participants Achieving a 100% Improvement From Baseline in Psoriasis Area and Severity Index (PASI) Score at Each Visit Through Week 24
Description: as for outcome 1
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Percentage of participants
  Week 2 | 0.0 [0.0 to 2.7] | 0.0 [0.0 to 2.7]
  Week 4 | 0.0 [0.0 to 2.7] | 0.7 [0.0 to 4.0]
  Week 8 | 0.0 [0.0 to 2.7] | 1.5 [0.2 to 5.2]
  Week 12 | 3.8 [1.2 to 8.6] | 2.2 [0.5 to 6.3]
  Week 16 | 7.5 [3.7 to 13.4] | 4.4 [1.6 to 9.3]
  Week 20 | 14.3 [8.8 to 21.4] | 7.3 [3.6 to 13.0]
  Week 24 | 14.3 [8.8 to 21.4] | 8.8 [4.6 to 14.8]
Statistical Analysis 1: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 2; Test type: Superiority or Other; The P-value at Week 2 was to be calculated by Fisher Exact method but was not estimable as the percentage of participants achieving 100% improvement in PASI in both treatment groups were 0%; Proportion difference = 0.00, 95% CI 2-sided [-0.74 to 0.74]
Statistical Analysis 2: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 4; Test type: Superiority or Other; p = 1.0000, Fisher Exact; Proportion difference = -0.73, 95% CI 2-sided [-2.90 to 1.44]
Statistical Analysis 3: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 8; Test type: Superiority or Other; p = 0.4983, Fisher Exact; Proportion difference = -1.46, 95% CI 2-sided [-4.21 to 1.29]
Statistical Analysis 4: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 12; Test type: Superiority or Other; p = 0.4957, Fisher Exact; Proportion difference = 1.57, 95% CI 2-sided [-3.23 to 6.37]
Statistical Analysis 5: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 16; Test type: Superiority or Other; p = 0.3115, Fisher Exact; Proportion difference = 3.14, 95% CI 2-sided [-3.24 to 9.52]
Statistical Analysis 6: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 20; Test type: Superiority or Other; p = 0.0773, Fisher Exact; Proportion difference = 6.99, 95% CI 2-sided [-1.13 to 15.10]
Statistical Analysis 7: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 24; Test type: Superiority or Other; p = 0.1830, Fisher Exact; Proportion difference = 5.53, 95% CI 2-sided [-2.82 to 13.87]

6. Secondary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) Score at Each Visit Through Week 24
Description: PASI: Combined assessment of lesion severity and area affected into single score; range: 0(no disease) to 72(maximal disease). Body was divided into 4 sections (head, arms, trunk, legs); each area scored by itself and scores were combined for final PASI. For each section, percent area of skin involved estimated: 0 (0%) to 6 (90 - 100%), and severity was estimated by clinical signs: erythema, induration, and desquamation; scale: 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each section * area score * weight of section (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4).
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on scale
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Units on scale
  Week 2 | -4.5 (0.4) | -3.2 (0.4)
  Week 4 | -8.7 (0.5) | -6.8 (0.4)
  Week 8 | -13.6 (0.5) | -10.6 (0.5)
  Week 12 | -16.2 (0.5) | -12.6 (0.5)
  Week 16 | -17.4 (0.5) | -14.6 (0.5)
  Week 20 | -17.5 (0.5) | -15.5 (0.5)
  Week 24 | -17.4 (0.5) | -15.4 (0.5)
Statistical Analysis 1: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 2; Test type: Superiority or Other; p = 0.0103, ANCOVA; ANCOVA model with treatment group as a factor and baseline measurement as a covariate were used for comparisons between treatment groups; Difference of adjusted mean change = -1.3, 95% CI 2-sided [-2.3 to -0.3]
Statistical Analysis 2: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 4; Test type: Superiority or Other; p = 0.0031, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -1.8, 95% CI 2-sided [-3.0 to -0.6]
Statistical Analysis 3: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 8; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -3.0, 95% CI 2-sided [-4.4 to -1.7]
Statistical Analysis 4: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -3.6, 95% CI 2-sided [-5.0 to -2.2]
Statistical Analysis 5: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 16; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -2.8, 95% CI 2-sided [-4.0 to -1.5]
Statistical Analysis 6: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 20; Test type: Superiority or Other; p = 0.0012, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -2.1, 95% CI 2-sided [-3.3 to -0.8]
Statistical Analysis 7: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 24; Test type: Superiority or Other; p = 0.0042, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -2.0, 95% CI 2-sided [-3.4 to -0.7]

7. Secondary Outcome: Time to Achieve Psoriasis Area and Severity Index (PASI) 50, PASI 75 and PASI 100 Over 24 Weeks
Description: Time taken to achieve first PASI was calculated using Kaplan-Meier estimate and presented as median. PASI 50=50% improvement from baseline in PASI; PASI 75=75% improvement from baseline in PASI; PASI 90=90% improvement from baseline in PASI; PASI 100=100% improvement from baseline in PASI. PASI score percent improvement =100*(baseline score - visit score)/baseline score.
Time Frame: Baseline to Week 24
Population: mITT population: all randomly assigned participants who received at least 1 ETN dose and had both baseline and on-therapy PASI evaluations. Observed cases (OC) analyses were performed including only those participants who were evaluated at the specified visits.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Days
  PASI 50 | 57 [56 to 57] | 57 [57 to 85]
  PASI 75 | 85 [84 to 85] | 113 [110 to 141]
  PASI 90 | 141 [113 to 170] | 171 [169 to NA] — Not estimable
  PASI 100 | NA [NA to NA] — Not estimable | NA [NA to NA] — Not estimable
Statistical Analysis 1: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison of treatment groups for PASI 50. Log rank test used to compare groups; CI based on product-limit method; Test type: Superiority or Other; p < 0.0001, Log Rank
Statistical Analysis 2: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison of treatment groups for PASI 75. Log rank test used to compare groups; CI based on product-limit method; Test type: Superiority or Other; p < 0.0001, Log Rank
Statistical Analysis 3: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison of treatment groups for PASI 90. Log rank test used to compare groups; CI based on product-limit method; Test type: Superiority or Other; p = 0.0053, Log Rank
Statistical Analysis 4: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison of treatment groups for PASI 100. Log rank test used to compare groups; CI based on product-limit method; Test type: Superiority or Other; p = 0.0432, Log Rank

8. Secondary Outcome: Percentage of Participants Achieving the Physician Global Assessment (PGA) of Psoriasis Responses of Clear (0) at Each Visit Through Week 24
Description: PGA of Psoriasis: score based on dermatologist's assessment of head, scalp, and neck psoriasis (averaged over all lesions). The PGA of Psoriasis scale ranges from 0 (no psoriasis) to 5 (severe disease). PGA score of 0 = Status of Clear.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Percentage of participants
  Week 2 | 0.0 [0.0 to 2.7] | 0.0 [0.0 to 2.7]
  Week 4 | 0.0 [0.0 to 2.7] | 0.7 [0.0 to 4.0]
  Week 8 | 1.5 [0.2 to 5.3] | 1.5 [0.2 to 5.2]
  Week 12 | 9.0 [4.7 to 15.2] | 2.9 [0.8 to 7.3]
  Week 16 | 12.8 [7.6 to 19.7] | 9.5 [5.1 to 15.7]
  Week 20 | 19.5 [13.2 to 27.3] | 10.9 [6.3 to 17.4]
  Week 24 | 21.1 [14.5 to 29.0] | 12.4 [7.4 to 19.1]
Statistical Analysis 1: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 2; Test type: Superiority or Other; Fisher Exact; Proportion difference = 0.00, 95% CI 2-sided [-0.74 to 0.74]
Statistical Analysis 2: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 4; Test type: Superiority or Other; p = 1.0000, Fisher Exact; Proportion difference = -0.73, 95% CI 2-sided [-2.90 to 1.44]
Statistical Analysis 3: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 8; Test type: Superiority or Other; p = 1.0000, Fisher Exact; Proportion difference = 0.04, 95% CI 2-sided [-3.58 to 3.67]
Statistical Analysis 4: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 12; Test type: Superiority or Other; p = 0.0401, Fisher Exact; Proportion difference = 6.10, 95% CI 2-sided [-0.26 to 12.47]
Statistical Analysis 5: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 16; Test type: Superiority or Other; p = 0.4415, Fisher Exact; Proportion difference = 3.29, 95% CI 2-sided [-4.95 to 11.54]
Statistical Analysis 6: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 20; Test type: Superiority or Other; p = 0.0617, Fisher Exact; Proportion difference = 8.60, 95% CI 2-sided [-0.67 to 17.87]
Statistical Analysis 7: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 24; Test type: Superiority or Other; p = 0.0720, Fisher Exact; Proportion difference = 8.64, 95% CI 2-sided [-0.96 to 18.24]

9. Secondary Outcome: Percentage of Participants Achieving the Physician Global Assessment (PGA) of Psoriasis Responses Clear/Almost Clear (0, 1) at Each Visit Through Week 24
Description: PGA of Psoriasis: score based on dermatologist's assessment of head, scalp, and neck psoriasis (averaged over all lesions). The PGA of Psoriasis scale ranges from 0 (no psoriasis) to 5 (severe disease). PGA score of 0 = Status of Clear; 1 = Almost Clear.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Percentage of participants
  Week 2 | 0.8 [0.0 to 4.1] | 2.2 [0.5 to 6.3]
  Week 4 | 12.8 [7.6 to 19.7] | 6.6 [3.0 to 12.1]
  Week 8 | 33.8 [25.9 to 42.5] | 18.2 [12.2 to 25.7]
  Week 12 | 54.9 [46.0 to 63.5] | 32.8 [25.1 to 41.4]
  Week 16 | 60.9 [52.1 to 69.2] | 47.4 [38.9 to 56.1]
  Week 20 | 65.4 [56.7 to 73.4] | 50.4 [41.7 to 59.0]
  Week 24 | 69.9 [61.4 to 77.6] | 50.4 [41.7 to 59.0]
Statistical Analysis 1: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 2; Test type: Superiority or Other; p = 0.6223, Fisher Exact; Proportion difference = -1.45, 95% CI 2-sided [-5.07 to 2.16]
Statistical Analysis 2: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 4; Test type: Superiority or Other; p = 0.1000, Fisher Exact; Proportion difference = 6.21, 95% CI 2-sided [-1.56 to 13.98]
Statistical Analysis 3: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 8; Test type: Superiority or Other; p = 0.0037, Fisher Exact; Proportion difference = 15.59, 95% CI 2-sided [4.53 to 26.65]
Statistical Analysis 4: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 12; Test type: Superiority or Other; p = 0.0004, Fisher Exact; Proportion difference = 22.04, 95% CI 2-sided [9.75 to 34.33]
Statistical Analysis 5: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 16; Test type: Superiority or Other; p = 0.0285, Fisher Exact; Proportion difference = 13.46, 95% CI 2-sided [0.94 to 25.97]
Statistical Analysis 6: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 20; Test type: Superiority or Other; p = 0.0139, Fisher Exact; Proportion difference = 15.05, 95% CI 2-sided [2.67 to 27.43]
Statistical Analysis 7: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 24; Test type: Superiority or Other; p = 0.0012, Fisher Exact; Proportion difference = 19.56, 95% CI 2-sided [7.38 to 31.74]

10. Secondary Outcome: Percentage of Participants Achieving the Physician Global Assessment (PGA) of Psoriasis Responses of Clear/Almost Clear/Mild (0, 1, 2) at Each Visit Through Week 24
Description: PGA of Psoriasis: score based on dermatologist's assessment of head, scalp, and neck psoriasis (averaged over all lesions). The PGA of Psoriasis scale ranges from 0 (no psoriasis) to 5 (severe disease). PGA score of 0 = Status of Clear; 1 = Almost Clear and 2 = Mild.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Percentage of participants
  Week 2 | 27.1 [19.7 to 35.5] | 22.1 [15.4 to 30.0]
  Week 4 | 46.6 [37.9 to 55.5] | 38.0 [29.8 to 46.6]
  Week 8 | 72.9 [64.5 to 80.3] | 59.1 [50.4 to 67.4]
  Week 12 | 88.7 [82.1 to 93.5] | 69.3 [60.9 to 76.9]
  Week 16 | 88.7 [82.1 to 93.5] | 75.2 [67.1 to 82.2]
  Week 20 | 88.7 [82.1 to 93.5] | 78.1 [70.2 to 84.7]
  Week 24 | 89.5 [83.0 to 94.1] | 78.1 [70.2 to 84.7]
Statistical Analysis 1: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 2; Test type: Superiority or Other; p = 0.3956, Fisher Exact; Proportion difference = 5.01, 95% CI 2-sided [-6.01 to 16.03]
Statistical Analysis 2: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 4; Test type: Superiority or Other; p = 0.1754, Fisher Exact; Proportion difference = 8.66, 95% CI 2-sided [-3.82 to 21.14]
Statistical Analysis 3: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 8; Test type: Superiority or Other; p = 0.0207, Fisher Exact; Proportion difference = 13.81, 95% CI 2-sided [1.90 to 25.72]
Statistical Analysis 4: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 12; Test type: Superiority or Other; p < 0.0001, Fisher Exact; Proportion difference = 19.38, 95% CI 2-sided [9.23 to 29.53]
Statistical Analysis 5: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 16; Test type: Superiority or Other; p = 0.0044, Fisher Exact; Proportion difference = 13.54, 95% CI 2-sided [3.79 to 23.29]
Statistical Analysis 6: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 20; Test type: Superiority or Other; p = 0.0223, Fisher Exact; Proportion difference = 10.62, 95% CI 2-sided [1.11 to 20.13]
Statistical Analysis 7: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 24; Test type: Superiority or Other; p = 0.0133, Fisher Exact; Proportion difference = 11.37, 95% CI 2-sided [1.96 to 20.78]

11. Secondary Outcome: Time to First Physician Global Assessment (PGA) of Psoriasis of Clear/Almost Clear (0, 1), or Clear/Almost Clear/Mild (0, 1, 2) Over 24 Weeks
Description: Time taken to achieve PGA was calculated using Kaplan-Meier estimate and presented as median. Assessment of clear or almost clear or Mild = PGA score of 0 (no evidence) or 1 (minimal/faint) or 2 (mild plaque elevation, mild fine scales predominates or light red coloration).
Time Frame: Baseline to Week 24
Population: mITT population: all randomly assigned participants who received at least 1 ETN dose and had both baseline and on-therapy PASI evaluations. OC analyses were performed including only those participants who were evaluated at the specified visits.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Days
  PGA Clear / Almost Clear (0, 1) | 85 [85 to 89] | 114 [112 to 167]
  PGA Clear / Almost Clear / Mild (0, 1, 2) | 53 [29 to 57] | 57 [56 to 57]
Statistical Analysis 1: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups for PGA Clear/Almost Clear (0,1). Log rank test used to compare groups; CI based on product-limit method; Test type: Superiority or Other; p = 0.0003, Log Rank
Statistical Analysis 2: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups for PGA Clear/Almost Clear/Mild (0,1,2). Log rank test used to compare groups; CI based on product-limit method; Test type: Superiority or Other; p = 0.0022, Log Rank

12. Secondary Outcome: Change From Baseline in Physician Global Assessment (PGA) of Psoriasis at Each Visit Through Week 24
Description: PGA of Psoriasis: score based on dermatologist's assessment of disease averaged over all lesions of head, scalp, and neck. Overall lesions were graded for induration, erythema, and scaling; range: 0 (no evidence) to 5 (severe). The sum of the 3 scores was divided by 3 to obtain a final PGA score. Higher scores indicate greater severity of disease.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on scale
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Units on scale
  Week 2 | -0.4 (0.0) | -0.3 (0.0)
  Week 4 | -0.9 (0.1) | -0.7 (0.1)
  Week 8 | -1.4 (0.1) | -1.1 (0.1)
  Week 12 | -1.9 (0.1) | -1.4 (0.1)
  Week 16 | -2.0 (0.1) | -1.7 (0.1)
  Week 20 | -2.1 (0.1) | -1.7 (0.1)
  Week 24 | -2.1 (0.1) | -1.8 (0.1)
Statistical Analysis 1: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 2; Test type: Superiority or Other; p = 0.0193, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -0.2, 95% CI 2-sided [-0.3 to -0.0]
Statistical Analysis 2: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 4; Test type: Superiority or Other; p = 0.0114, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -0.2, 95% CI 2-sided [-0.4 to -0.1]
Statistical Analysis 3: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 8; Test type: Superiority or Other; p = 0.0006, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -0.3, 95% CI 2-sided [-0.5 to -0.2]
Statistical Analysis 4: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -0.5, 95% CI 2-sided [-0.7 to -0.3]
Statistical Analysis 5: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 16; Test type: Superiority or Other; p = 0.0058, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -0.3, 95% CI 2-sided [-0.5 to -0.1]
Statistical Analysis 6: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 20; Test type: Superiority or Other; p = 0.0018, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -0.4, 95% CI 2-sided [-0.6 to -0.1]
Statistical Analysis 7: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 24; Test type: Superiority or Other; p = 0.0009, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -0.4, 95% CI 2-sided [-0.6 to -0.2]

13. Other Pre Specified Outcome: Change From Baseline in Subject Global Assessment (SGA) of Itching at Each Visit Through Week 24
Description: SGA of Psoriasis: score based on participant's assessment of itching at a scale of 0 to 5; where 0 = no itching and 5 = severe itching.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on scale
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Units on scale
  Week 2 | -0.8 (0.1) | -0.7 (0.1)
  Week 4 | -1.5 (0.1) | -1.1 (0.1)
  Week 8 | -2.0 (0.1) | -1.4 (0.1)
  Week 12 | -2.4 (0.1) | -1.6 (0.1)
  Week 16 | -2.2 (0.1) | -1.8 (0.1)
  Week 20 | -2.3 (0.1) | -1.8 (0.1)
  Week 24 | -2.2 (0.1) | -2.0 (0.1)
Statistical Analysis 1: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 2; Test type: Superiority or Other; p = 0.6396, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -0.1, 95% CI 2-sided [-0.3 to 0.2]
Statistical Analysis 2: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 4; Test type: Superiority or Other; p = 0.0074, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -0.4, 95% CI 2-sided [-0.7 to -0.1]
Statistical Analysis 3: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 8; Test type: Superiority or Other; p = 0.0007, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -0.6, 95% CI 2-sided [-0.9 to -0.2]
Statistical Analysis 4: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -0.8, 95% CI 2-sided [-1.1 to -0.5]
Statistical Analysis 5: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 16; Test type: Superiority or Other; p = 0.0040, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -0.5, 95% CI 2-sided [-0.8 to -0.1]
Statistical Analysis 6: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 20; Test type: Superiority or Other; p = 0.0004, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -0.6, 95% CI 2-sided [-0.9 to -0.3]
Statistical Analysis 7: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 24; Test type: Superiority or Other; p = 0.1799, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -0.2, 95% CI 2-sided [-0.5 to -0.1]

14. Other Pre Specified Outcome: Change From Baseline in Subject Global Assessment (SGA) of Joint Pain at Each Visit Through Week 24
Description: SGA of Joint Pain: score based on participant's assessment of joint pain at a scale of 0 to 5; where 0 = no pain and 5 = severe pain.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on scale
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Units on scale
  Week 2 | -0.4 (0.1) | -0.5 (0.1)
  Week 4 | -0.7 (0.1) | -0.5 (0.1)
  Week 8 | -0.7 (0.1) | -0.6 (0.1)
  Week 12 | -0.8 (0.1) | -0.6 (0.1)
  Week 16 | -0.8 (0.1) | -0.6 (0.1)
  Week 20 | -0.9 (0.1) | -0.6 (0.1)
  Week 24 | -0.8 (0.1) | -0.8 (0.1)
Statistical Analysis 1: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 2; Test type: Superiority or Other; p = 0.7757, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = 0.0, 95% CI 2-sided [-0.2 to 0.3]
Statistical Analysis 2: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 4; Test type: Superiority or Other; p = 0.2112, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -0.2, 95% CI 2-sided [-0.4 to 0.1]
Statistical Analysis 3: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 8; Test type: Superiority or Other; p = 0.5467, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -0.1, 95% CI 2-sided [-0.3 to 0.2]
Statistical Analysis 4: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 12; Test type: Superiority or Other; p = 0.3684, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -0.1, 95% CI 2-sided [-0.4 to 0.1]
Statistical Analysis 5: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 16; Test type: Superiority or Other; p = -0.2046, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -0.2, 95% CI 2-sided [-0.4 to 0.1]
Statistical Analysis 6: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 20; Test type: Superiority or Other; p = 0.0649, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -0.2, 95% CI 2-sided [-0.5 to 0.0]
Statistical Analysis 7: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 24; Test type: Superiority or Other; p = 0.8683, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -0.0, 95% CI 2-sided [-0.3 to 0.2]

15. Other Pre Specified Outcome: Change From Baseline in Subject Global Assessment (SGA) of Psoriasis at Each Visit Through Week 24
Description: SGA of Psoriasis: score based on participant's assessment of psoriasis disease activity at a scale of 0 to 5; where 0 = good and 5 = severe.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on scale
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Units on scale
  Week 2 | -1.0 (0.1) | -1.0 (0.1)
  Week 4 | -1.8 (0.1) | -1.4 (0.1)
  Week 8 | -2.1 (0.1) | -1.7 (0.1)
  Week 12 | -2.5 (0.1) | -1.9 (0.1)
  Week 16 | -2.6 (0.1) | -2.0 (0.1)
  Week 20 | -2.6 (0.1) | -2.1 (0.1)
  Week 24 | -2.5 (0.1) | -2.2 (0.1)
Statistical Analysis 1: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 2; Test type: Superiority or Other; p = 0.8898, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -0.0, 95% CI 2-sided [-0.3 to 0.2]
Statistical Analysis 2: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 4; Test type: Superiority or Other; p = 0.0090, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -0.4, 95% CI 2-sided [-0.7 to -0.1]
Statistical Analysis 3: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 8; Test type: Superiority or Other; p = 0.0028, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -0.4, 95% CI 2-sided [-0.7 to -0.2]
Statistical Analysis 4: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 12; Test type: Superiority or Other; p = 0.0001, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -0.6, 95% CI 2-sided [-0.9 to -0.3]
Statistical Analysis 5: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 16; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -0.6, 95% CI 2-sided [-0.9 to -0.3]
Statistical Analysis 6: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 20; Test type: Superiority or Other; p = 0.0016, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -0.5, 95% CI 2-sided [-0.8 to -0.2]
Statistical Analysis 7: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 24; Test type: Superiority or Other; p = 0.0602, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -0.3, 95% CI 2-sided [-0.6 to 0.0]

16. Secondary Outcome: Change From Baseline in Percent Body Surface Area (BSA) Involvement of Psoriasis at Each Visit Through Week 24
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of BSA
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Percentage of BSA
  Week 2 | -1.8 (7.0) | -0.3 (6.7)
  Week 4 | -5.3 (10.1) | -3.1 (7.7)
  Week 8 | -13.4 (15.2) | -8.4 (11.8)
  Week 12 | -20.0 (19.2) | -12.7 (15.7)
  Week 16 | -23.8 (19.7) | -15.9 (15.9)
  Week 20 | -25.4 (18.8) | -18.2 (16.3)
  Week 24 | -25.9 (19.2) | -19.0 (17.2)

17. Secondary Outcome: Change From Baseline in the Photographed Image of Lesions in Selected Participants
Description: Compare the before and after photographs with the clinical assessments (Psoriasis Area and Severity Index, Physician's Global Assessment) taken at the same time for illustration purposes. Measured as yes or no for change.
Time Frame: Baseline to Week 24
Population: The data was not collected as planned.
Measure: Number; unit: Units on scale
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Percentage of Participants Not Using Topical Preparations at Each Visit From Week 12 Through Week 24
Description: Moderate topical steroids to very potent topical steroids, topical vitamin D analogs, topical steroids in combination with vitamin D analogs, and anthralin compounds were prohibited for 14 days before the baseline visit until week 12.
Time Frame: From Week 12 to Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Percentage of participants
  Week 12 | 89.5 | 89.1
  Week 16 | 85.0 | 81.0
  Week 20 | 86.5 | 82.5
  Week 24 | 85.7 | 83.2
Statistical Analysis 1: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 12; Test type: Superiority or Other; p = 1.0000, Fisher Exact; Proportion difference = 0.42, 95% CI 2-sided [-7.70 to 8.55]
Statistical Analysis 2: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 16; Test type: Superiority or Other; p = 0.4213, Fisher Exact; Proportion difference = 3.94, 95% CI 2-sided [-5.75 to 13.63]
Statistical Analysis 3: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 20; Test type: Superiority or Other; p = 0.4039, Fisher Exact; Proportion difference = 3.98, 95% CI 2-sided [-5.38 to 13.35]
Statistical Analysis 4: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 24; Test type: Superiority or Other; p = 0.6168, Fisher Exact; Proportion difference = 2.50, 95% CI 2-sided [-6.87 to 11.88]

19. Other Pre Specified Outcome: Change From Baseline in Psoriatic Arthritis Screening and Evaluation (PASE) Total Score at Week 12
Description: PASE a participant-administered questionnaire and a simple scoring system to assist physicians in screening participants with psoriasis for evidence of psoriatic arthritis with two sub-scales: system sub-scale and function sub-scale. Total of 15 questions in both sub-scales (7 questions in system and 8 in function sub-scale) to score from 1 to 5; where 1 = strongly disagree and 5 = strongly agree. The total of system and function scores provides the total PASE score ranging from 15 to 75 where higher scores indicate greater severity.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on scale
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 129 | 133
Units on scale | -3.7 (1.0) | -3.5 (0.9)
Statistical Analysis 1: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Test type: Superiority or Other; p = 0.8620, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -0.2, 95% CI 2-sided [-2.8 to 2.3]

20. Other Pre Specified Outcome: Percentage of Participants Evaluated Using Psoriasis Physician Satisfaction Questionnaire (PPSQ): Consider Patient's Condition Satisfactory From Baseline at Each Visit Through Week 24
Description: Physician Psoriasis Satisfaction Questionnaire (PPSQ) included two global satisfaction questions to which physicians respond either 'satisfactory' or 'not satisfactory.' These are: 1) whether the participant's current condition is satisfactory, considering psoriasis symptoms, skin appearance and all other problems that psoriasis causes; 2) whether the participant's current primary psoriasis therapy is satisfactory, considering psoriasis symptoms, skin appearance, therapy side effects and therapy ease/difficulty of use. Each of these questions was summarized for change from baseline.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Percentage of participants
  Week 2 | 33.1 [25.2 to 41.8] | 27.4 [20.1 to 35.7]
  Week 4 | 53.4 [44.5 to 62.1] | 38.7 [30.5 to 47.4]
  Week 8 | 68.4 [59.8 to 76.2] | 54.0 [45.3 to 62.6]
  Week 12 | 87.2 [80.3 to 92.4] | 65.7 [57.1 to 73.6]
  Week 16 | 85.7 [78.6 to 91.2] | 75.2 [67.1 to 82.2]
  Week 20 | 87.2 [80.3 to 92.4] | 75.2 [67.1 to 82.2]
  Week 24 | 86.5 [79.5 to 91.8] | 75.2 [67.1 to 82.2]
Statistical Analysis 1: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 2; Test type: Superiority or Other; p = 0.3525, Fisher Exact; Proportion difference = 5.68, 95% CI 2-sided [-6.05 to 17.40]
Statistical Analysis 2: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 4; Test type: Superiority or Other; p = 0.0202, Fisher Exact; Proportion difference = 14.70, 95% CI 2-sided [2.19 to 27.20]
Statistical Analysis 3: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 8; Test type: Superiority or Other; p = 0.0178, Fisher Exact; Proportion difference = 14.41, 95% CI 2-sided [2.17 to 26.64]
Statistical Analysis 4: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 12; Test type: Superiority or Other; p < 0.0001, Fisher Exact; Proportion difference = 21.52, 95% CI 2-sided [11.02 to 32.03]
Statistical Analysis 5: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 16; Test type: Superiority or Other; p = 0.0325, Fisher Exact; Proportion difference = 10.53, 95% CI 2-sided [0.43 to 20.64]
Statistical Analysis 6: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 20; Test type: Superiority or Other; p = 0.0129, Fisher Exact; Proportion difference = 12.04, 95% CI 2-sided [2.10 to 21.97]
Statistical Analysis 7: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 24; Test type: Superiority or Other; p = 0.0209, Fisher Exact; Proportion difference = 11.28, 95% CI 2-sided [1.26 to 21.30]

21. Other Pre Specified Outcome: Percentage of Participants Evaluated by Physicians Using Psoriasis Physician Satisfaction Questionnaire (PPSQ): Consider Primary Psoriasis Therapy Satisfactory From Baseline at Each Visit Through Week 24
Description: Physician Psoriasis Satisfaction Questionnaire (PPSQ) includes two global satisfaction questions to which physicians respond either 'satisfactory' or 'not satisfactory.' These are: 1) whether the participant's current condition is satisfactory, considering psoriasis symptoms, skin appearance and all other problems that psoriasis causes; 2) whether the participant's current primary psoriasis therapy is satisfactory, considering psoriasis symptoms, skin appearance, therapy side effects and therapy ease/difficulty of use. Each of these questions was summarized for change from baseline.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Percentage of participants
  Week 2 | 66.9 [58.2 to 74.8] | 54.8 [46.0 to 63.4]
  Week 4 | 77.4 [69.4 to 84.2] | 68.6 [60.1 to 76.3]
  Week 8 | 83.5 [76.0 to 89.3] | 72.3 [64.0 to 79.6]
  Week 12 | 91.7 [85.7 to 95.8] | 83.2 [75.9 to 89.0]
  Week 16 | 91.7 [85.7 to 95.8] | 84.7 [77.5 to 90.3]
  Week 20 | 91.7 [85.7 to 95.8] | 83.9 [76.7 to 89.7]
  Week 24 | 88.7 [82.1 to 93.5] | 81.0 [73.4 to 87.2]
Statistical Analysis 1: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 2; Test type: Superiority or Other; p = 0.0461, Fisher Exact; Proportion difference = 12.10, 95% CI 2-sided [-0.24 to 24.44]
Statistical Analysis 2: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 4; Test type: Superiority or Other; p = 0.1314, Fisher Exact; Proportion difference = 8.83, 95% CI 2-sided [-2.44 to 20.10]
Statistical Analysis 3: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 8; Test type: Superiority or Other; p = 0.0289, Fisher Exact; Proportion difference = 11.20, 95% CI 2-sided [0.65 to 21.74]
Statistical Analysis 4: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 12; Test type: Superiority or Other; p = 0.0433, Fisher Exact; Proportion difference = 8.52, 95% CI 2-sided [-0.04 to 17.07]
Statistical Analysis 5: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 16; Test type: Superiority or Other; p = 0.0902, Fisher Exact; Proportion difference = 7.06, 95% CI 2-sided [-1.32 to 15.43]
Statistical Analysis 6: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 20; Test type: Superiority or Other; p = 0.0630, Fisher Exact; Proportion difference = 7.79, 95% CI 2-sided [-0.68 to 16.26]
Statistical Analysis 7: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 24; Test type: Superiority or Other; p = 0.0907, Fisher Exact; Proportion difference = 7.70, 95% CI 2-sided [-1.53 to 16.93]

22. Secondary Outcome: Mean Psoriasis Subject Satisfaction Questionnaire (PSSQ) Scores at Week 12
Description: PSSQ: participant's assessment that includes 18 items, 16 items (1-16) scored using Likert score with scores from 0 (very dissatisfied) to 4 (very satisfied) and 5 ( never had this problem). Only those participants who do not have score of 5 at baseline included in the item 1-16 analyses. Two items (17, 18) are with Yes/No answers. The scores of items 1-16 for change from baseline are summarized here.
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Units on scale
  Overall appearance of your skin | 3.2 (0.9) | 2.6 (1.2)
  Flaking skin | 3.3 (1.0) | 2.7 (1.2)
  Skin redness | 3.2 (1.0) | 2.5 (1.2)
  Skin tightness | 3.4 (1.1) | 3.0 (1.2)
  Skin bleeding | 3.8 (1.0) | 3.2 (1.3)
  Burning sensation in the skin | 3.8 (1.1) | 3.0 (1.4)
  Skin pain | 3.8 (1.1) | 3.1 (1.4)
  Joint pain | 3.1 (1.3) | 2.9 (1.4)
  Comfort level with your appearance | 3.2 (1.0) | 2.7 (1.2)
  Anxiety | 3.2 (1.3) | 3.1 (1.3)
  Depression | 3.5 (1.3) | 3.2 (1.4)
  Fatigue | 3.0 (1.1) | 2.9 (1.2)
  How others respond to your appearance | 3.5 (1.1) | 2.9 (1.3)
  How your skin affects social, leisure activities | 3.1 (1.2) | 2.7 (1.4)
  Satisfaction with psoriasis treatment in general | 3.3 (0.8) | 2.9 (1.0)
  Would like to continue with my current treatment | 3.7 (0.6) | 3.5 (0.9)

23. Secondary Outcome: Mean Psoriasis Subject Satisfaction Questionnaire (PSSQ) Scores at Week 24
Description: PSSQ: participant's assessment that includes 18 items, 16 items (1-16) scored using Likert score with scores from 0 (very dissatisfied) to 4 (very satisfied) and 5 (never had this problem). Only those participants who do not have score of 5 at baseline included in the item 1-16 analyses. Two items (17, 18) are with Yes/No answers. The scores of items 1-16 for change from baseline are summarized here.
Time Frame: Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Units on scale
  Overall appearance of your skin | 3.2 (1.0) | 2.8 (1.2)
  Flaking skin | 3.4 (1.1) | 3.0 (1.3)
  Skin redness | 3.3 (1.1) | 2.9 (1.3)
  Skin tightness | 3.5 (1.1) | 3.2 (1.3)
  Skin bleeding | 3.8 (1.1) | 3.3 (1.4)
  Burning sensation in the skin | 3.7 (1.1) | 3.3 (1.4)
  Skin pain | 3.7 (1.1) | 3.3 (1.4)
  Joint pain | 3.3 (1.2) | 3.1 (1.5)
  Comfort level with your appearance | 3.2 (1.0) | 2.9 (1.2)
  Anxiety | 3.4 (1.2) | 3.2 (1.5)
  Depression | 3.3 (1.3) | 3.4 (1.4)
  Fatigue | 3.1 (1.1) | 3.0 (1.3)
  How others respond to your appearance | 3.4 (1.0) | 3.2 (1.2)
  How your skin affects social, leisure activities | 3.4 (1.0) | 3.2 (1.4)
  Satisfaction with psoriasis treatment in general | 3.2 (1.0) | 3.1 (1.0)
  Would like to continue with my current treatment | 3.5 (1.0) | 3.4 (1.0)

24. Other Pre Specified Outcome: Percentage of Participants Who Were Considered Satisfied With Health State According to Psoriasis Subject Satisfaction Questionnaire (PSSQ)
Description: PSSQ: participant's assessment that includes 18 items, 16 items (1-16) scored using Likert score with scores from 0 (very dissatisfied) to 4 (very satisfied) and 5 (never had this problem). Only those participants who do not have score of 5 at baseline included in the item 1-16 analyses. Two items (17, 18) with Yes/No answers are summarized here.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Percentage of participants
  Week 2 | 47.4 [38.7 to 56.2] | 44.1 [35.6 to 52.9]
  Week 4 | 68.4 [59.8 to 76.2] | 59.1 [50.4 to 67.4]
  Week 8 | 81.2 [73.5 to 87.5] | 69.3 [60.9 to 76.9]
  Week 12 | 85.0 [77.7 to 90.6] | 70.8 [62.4 to 78.3]
  Week 16 | 85.7 [78.6 to 91.2] | 73.7 [65.5 to 80.9]
  Week 20 | 85.0 [77.7 to 90.6] | 75.9 [67.9 to 82.8]
  Week 24 | 85.0 [77.7 to 90.6] | 74.5 [66.3 to 81.5]
Statistical Analysis 1: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 2; Test type: Superiority or Other; p = 0.6255, Fisher Exact; Proportion difference = 3.25, 95% CI 2-sided [-9.39 to 15.90]
Statistical Analysis 2: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 4; Test type: Superiority or Other; p = 0.1292, Fisher Exact; Proportion difference = 9.30, 95% CI 2-sided [-2.85 to 21.45]
Statistical Analysis 3: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 8; Test type: Superiority or Other; p = 0.0251, Fisher Exact; Proportion difference = 11.86, 95% CI 2-sided [0.94 to 22.78]
Statistical Analysis 4: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 12; Test type: Superiority or Other; p = 0.0055, Fisher Exact; Proportion difference = 14.16, 95% CI 2-sided [3.68 to 24.64]
Statistical Analysis 5: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 16; Test type: Superiority or Other; p = 0.0159, Fisher Exact; Proportion difference = 11.99, 95% CI 2-sided [1.78 to 22.20]
Statistical Analysis 6: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 20; Test type: Superiority or Other; p = 0.0672, Fisher Exact; Proportion difference = 9.05, 95% CI 2-sided [-1.08 to 19.18]
Statistical Analysis 7: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 24; Test type: Superiority or Other; p = 0.0351, Fisher Exact; Proportion difference = 10.51, 95% CI 2-sided [0.27 to 20.75]

25. Other Pre Specified Outcome: Percentage of Participants Who Were Considered Satisfied With Primary Psoriasis Treatment According to Psoriasis Subject Satisfaction Questionnaire (PSSQ)
Description: as for outcome 24
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Percentage of participants
  Week 2 | 82.7 | 76.5
  Week 4 | 88.0 | 82.5
  Week 8 | 92.5 | 82.5
  Week 12 | 92.5 | 82.5
  Week 16 | 91.0 | 86.1
  Week 20 | 91.7 | 86.1
  Week 24 | 87.2 | 83.2
Statistical Analysis 1: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 2; Test type: Superiority or Other; p = 0.2283, Fisher Exact; Proportion difference = 6.24, 95% CI 2-sided [-4.11 to 16.58]
Statistical Analysis 2: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 4; Test type: Superiority or Other; p = 0.2326, Fisher Exact; Proportion difference = 5.49, 95% CI 2-sided [-3.68 to 14.66]
Statistical Analysis 3: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 8; Test type: Superiority or Other; p = 0.0165, Fisher Exact; Proportion difference = 10.00, 95% CI 2-sided [1.47 to 18.52]
Statistical Analysis 4: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 12; Test type: Superiority or Other; p = 0.0165, Fisher Exact; Proportion difference = 10.00, 95% CI 2-sided [1.47 to 18.52]
Statistical Analysis 5: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 16; Test type: Superiority or Other; p = 0.2536, Fisher Exact; Proportion difference = 4.85, 95% CI 2-sided [-3.46 to 13.15]
Statistical Analysis 6: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 20; Test type: Superiority or Other; p = 0.1761, Fisher Exact; Proportion difference = 5.60, 95% CI 2-sided [-2.59 to 13.78]
Statistical Analysis 7: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 24; Test type: Superiority or Other; p = 0.3943, Fisher Exact; Proportion difference = 4.01, 95% CI 2-sided [-5.18 to 13.20]

26. Other Pre Specified Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score to Week 24
Description: DLQI is the dermatology-specific quality of life measure used for psoriatic population. The 10-item questionnaire has a score range of 0 to 30 with higher scores indicating poor quality of life. An estimate of the minimal clinically important difference of the DLQI total score is a 5 point improvement. Total score range: 0 (best) to 30 (worst).
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on scale
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Units on scale
  Week 2 | -4.6 (0.4) | -4.3 (0.4)
  Week 4 | -7.1 (0.5) | -5.9 (0.4)
  Week 8 | -9.0 (0.5) | -7.0 (0.5)
  Week 12 | -10.2 (0.5) | -8.1 (0.5)
  Week 16 | -10.7 (0.4) | -8.8 (0.4)
  Week 20 | -10.5 (0.5) | -9.0 (0.5)
  Week 24 | -10.5 (0.5) | -9.2 (0.5)
Statistical Analysis 1: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 2; Test type: Superiority or Other; p = 0.5748, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -0.3, 95% CI 2-sided [-1.5 to 0.8]
Statistical Analysis 2: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 4; Test type: Superiority or Other; p = 0.0471, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -1.2, 95% CI 2-sided [-2.4 to -0.0]
Statistical Analysis 3: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 8; Test type: Superiority or Other; p = 0.0025, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -2.0, 95% CI 2-sided [-3.3 to -0.7]
Statistical Analysis 4: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 12; Test type: Superiority or Other; p = 0.0009, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -2.2, 95% CI 2-sided [-3.5 to -0.9]
Statistical Analysis 5: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 16; Test type: Superiority or Other; p = 0.0015, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -1.9, 95% CI 2-sided [-3.1 to -0.7]
Statistical Analysis 6: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 20; Test type: Superiority or Other; p = 0.0197, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -1.5, 95% CI 2-sided [-2.7 to -0.2]
Statistical Analysis 7: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 24; Test type: Superiority or Other; p = 0.0506, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -1.3, 95% CI 2-sided [-2.6 to 0.0]

27. Other Pre Specified Outcome: Change From Baseline in the Euro Quality of Life 5 Dimension (EQ-5D) Utility Index
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state (example "confined to bed"). Scoring formula developed by EuroQol Group assigns utility value for each domain in the profile. Score is transformed and results in total score range -0.594 to 1.000; higher score indicates better health state.
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on scale
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 130 | 134
Units on scale
  Week 12 | 0.21 (0.02) | 0.17 (0.02)
  Week 24 | 0.21 (0.02) | 0.15 (0.02)
Statistical Analysis 1: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 12; Test type: Superiority or Other; p = 0.0435, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = 0.04, 95% CI 2-sided [0.00 to 0.09]
Statistical Analysis 2: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 24; Test type: Superiority or Other; p = 0.0275, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = 0.05, 95% CI 2-sided [0.01 to 0.10]

28. Other Pre Specified Outcome: Change From Baseline in the Hospital Anxiety and Depression Scale (HADS) - Anxiety Score
Description: HADS: participant rated questionnaire with 2 subscales. HADS-A assesses state of generalized anxiety (anxious mood, restlessness, anxious thoughts, panic attacks); HADS-D assesses state of lost interest and diminished pleasure response (lowering of hedonic tone). Each subscale comprised of 7 items with range 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). Total score 0 to 21 for each subscale; higher score indicates greater severity of anxiety and depression symptoms.
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on scale
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 131 | 135
Units on scale
  Week 12 | -1.6 (0.3) | -1.6 (0.3)
  Week 24 | -1.9 (0.3) | -1.8 (0.3)
Statistical Analysis 1: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 12; Test type: Superiority or Other; p = 0.9473, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = 0.0, 95% CI 2-sided [-0.7 to 0.7]
Statistical Analysis 2: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 24; Test type: Superiority or Other; p = 0.8217, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of adjusted mean change = -0.1, 95% CI 2-sided [-0.8 to 0.6]

29. Other Pre Specified Outcome: Change From Baseline in the Hospital Anxiety and Depression Scale (HADS) - Depression Score
Description: as for outcome 28
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on scale
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 131 | 135
Units on scale
  Week 12 | -1.9 (0.3) | -1.3 (0.3)
  Week 24 | -2.2 (0.3) | -1.7 (0.3)
Statistical Analysis 1: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 12; Test type: Superiority or Other; p = 0.0539, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of Adjusted Mean Change = -0.7, 95% CI 2-sided [-1.4 to 0.0]
Statistical Analysis 2: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 24; Test type: Superiority or Other; p = 0.1494, ANCOVA; [statistical method as in outcome 6, analysis 1]; Difference of Adjusted Mean Change = -0.5, 95% CI 2-sided [-1.3 to 0.2]

30. Other Pre Specified Outcome: Work Productivity and Activity Impairment: Psoriasis (WPAI:PSO) at Week 12
Description: WPAI:PSO - participant rated questionnaire to assess effect of psoriasis on ability to work and perform regular activities in 4 areas: percent activity impairment (0 [no effect on daily activities] to 100 [psoriasis completely prevented from doing daily activities]), percent impairment while working (0 [no effect] to 100 [completely prevented from working]); percent work time missed due to psoriasis, and percent overall work impairment (0 [no effect] to 100 [completely prevented from working]).
Time Frame: Week 12
Population: mITT population: all randomized participants who received at least 1 ETN dose and had both baseline and on-therapy PASI evaluations. If participant had missing values at any time point, LOCF method of imputation used. 'n' signifies participants evaluated for this measure at each timepoint, for each group respectively.
Measure: Mean (Standard Deviation); unit: Percentage of indicated parameter
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 131 | 135
Percentage of indicated parameter
  Percent Activity Impairment (n=131, 135) | 16.87 (21.49) | 21.78 (25.65)
  Percent Impairment While Working (n=66, 78) | 10.25 (14.41) | 13.19 (20.43)
  Percent Overall Work Impairment (n=64, 71)) | 14.30 (21.49) | 16.88 (25.24)
  Percent Work Time Missed (n=66, 73) | 4.35 (16.86) | 4.85 (19.11)

31. Other Pre Specified Outcome: Work Productivity and Activity Impairment: Psoriasis (WPAI:PSO) at Week 24
Description: as for outcome 30
Time Frame: Week 24
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: Percentage of indicated parameter
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 131 | 135
Percentage of indicated parameter
  Percent Activity Impairment (n=131, 135)) | 13.28 (18.99) | 18.85 (24.58)
  Percent Impairment While Working (n=72, 81) | 8.00 (11.34) | 13.43 (19.57)
  Percent Overall Work Impairment (n=70, 76) | 12.78 (20.27) | 15.96 (23.05)
  Percent Work Time Missed (n=72, 78) | 5.03 (17.57) | 3.10 (13.91)

32. Other Pre Specified Outcome: Mean Medical Outcomes Study (MOS) Sleep Scale Scores at Week 12
Description: MOS scale has 12 questions to assess sleep quality & quantity: 1)time to fall asleep, 2)hours of sleep/night in past 4 weeks,3)sleep not peaceful, 4)got enough sleep to feel rested in morning,5)awaken short of breath/headache 6)feel drowsy in day,7)trouble going to sleep, 8)wake up during sleep; trouble going back to sleep,9)trouble staying awake in day, 10)Snoring,11)take naps in day,12)get amount of sleep needed. Sleep problem index(SPI) I:mean of 4,5,7,8,9,12; SPI II:mean of 1,3,4,5,6,7,8,9,12. All reported responses are on scale:0-100, higher scores indicate greater intensity of attribute.
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Units on scale
  Sleep Snoring | 35.7 (27.8) | 45.3 (30.3)
  Sleep Somnolence | 27.3 (19.8) | 28.8 (20.3)
  Sleep Short of Breath or Headache | 13.6 (20.8) | 15.3 (21.2)
  Sleep Adequacy | 59.8 (26.4) | 55.6 (24.4)
  Sleep Disturbance | 30.1 (21.3) | 28.4 (21.1)
  Sleep Quantity | 7.2 (1.4) | 6.9 (1.2)
  Sleep Problem Index I | 29.3 (17.8) | 30.4 (17.8)
  Sleep Problem Index II | 30.1 (17.5) | 30.8 (17.7)

33. Other Pre Specified Outcome: Mean Medical Outcomes Study (MOS) Sleep Scale Scores at Week 24
Description: MOS: participant rated questionnaire to assess sleep quality and quantity. Consists of a 9-item overall sleep problems index (length of time to fall asleep, how many hours of sleep each night during past 4 weeks); 7 subscales rated 1 (all the time) to 6 (none of the time): sleep disturbance, snoring, awaken short of breath (SOB) or with headache, somnolence adequacy, and sleep quantity. Scores are transformed (actual raw score minus lowest possible score divided by possible raw score range multiplied by 100); total score range = 0 to 100; higher score indicates greater intensity of attribute.
Time Frame: Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Units on scale
  Sleep Snoring | 38.2 (31.1) | 44.0 (31.3)
  Sleep Somnolence | 27.0 (18.4) | 28.1 (20.3)
  Sleep Short of Breath or Headache | 11.9 (17.3) | 13.9 (19.7)
  Sleep Adequacy | 59.8 (25.4) | 60.9 (26.7)
  Sleep Disturbance | 26.7 (19.8) | 26.6 (21.1)
  Sleep Quantity | 7.2 (1.5) | 7.0 (1.3)
  Sleep Problem Index I | 27.3 (15.9) | 27.7 (17.7)
  Sleep Problem Index II | 28.2 (15.7) | 28.4 (17.5)

34. Other Pre Specified Outcome: Mean Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Questionnaire Total Scores
Description: FACIT Fatigue questionnaire: Participant rated 13 items questionnaire to assess fatigue. For each question, participant rates his / her condition for the past week on a 5-point Likert scale ranging from 0 (not at all) to 4 (very much). Higher scores always represent less fatigue. The total FACIT-Fatigue score ranges from 0 to 52 and is the sum of non-missing item scores; divided by the number of non-missing items, then multiplied by 13. If more than 6 items were missing, the total score was missing.
Time Frame: Week 12 and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Units on scale
  Week 12 | 41.8 (8.1) | 40.1 (8.6)
  Week 24 | 41.9 (8.3) | 40.8 (9.1)

35. Other Pre Specified Outcome: Percentage of Participants With Emergency Room Visits
Description: As a part of pharmacoeconomic questionnaire, the visits to emergency room were evaluated and presented as Yes or No.
Time Frame: Week 12 and Week 24
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Percentage of participants
  Week 12 | 0.8 | 3.7
  Week 24 | 1.6 | 0.8
Statistical Analysis 1: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 12; Test type: Superiority or Other; p = 0.2139, Fisher Exact
Statistical Analysis 2: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 24; Test type: Superiority or Other; p = 1.0000, Fisher Exact

36. Other Pre Specified Outcome: Mean Number of Emergency Room Days
Description: As a part of pharmacoeconomic questionnaire, mean number of emergency room days were summarized.
Time Frame: Week 12 and Week 24
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Days
  Week 12 | 1.0 (NA) — Not estimable due to small sample size. | 3.6 (5.81)
  Week 24 | 1.0 (0.00) | 1.0 (NA) — Not estimable due to small sample size.

37. Other Pre Specified Outcome: Percentage of Participants With Doctor Visits
Description: As a part of pharmacoeconomic questionnaire, the percentage of participants who had doctor visits were presented as Yes or No.
Time Frame: Week 12 and Week 24
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Percentage of participants
  Week 12 | 29.8 | 36.8
  Week 24 | 31.7 | 31.7
Statistical Analysis 1: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 12; Test type: Superiority or Other; p = 0.2443, Fisher Exact
Statistical Analysis 2: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison between treatment groups at Week 24; Test type: Superiority or Other; p = 1.0000, Fisher Exact

38. Other Pre Specified Outcome: Mean Number of Doctor Visits
Description: As a part of pharmacoeconomic questionnaire, the mean number of doctor visits were summarized.
Time Frame: Week 12 and Week 24
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Visits
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Number analyzed (Participants) | 133 | 137
Visits
  Week 12 | 2.2 (1.25) | 3.3 (3.89)
  Week 24 | 2.4 (1.99) | 1.9 (1.28)
Statistical Analysis 1: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison of treatment groups at Week 12; Test type: Superiority or Other; p = 0.0807, ANCOVA
Statistical Analysis 2: Comparison: ETN 50 mg BW/QW vs ETN 50 mg QW/QW; Comparison of treatment groups at Week 24; Test type: Superiority or Other; p = 0.1454, ANCOVA

ADVERSE EVENTS:
Description: The same event may appear as both an Adverse Event and a Serious Adverse Event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | ETN 50 mg BW/QW | ETN 50 mg QW/QW
Serious Adverse Events (participants affected / at risk) | 3/136 | 4/137
Other Adverse Events (participants affected / at risk) | 97/136 | 91/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ETN 50 mg BW/QW (N=136) | ETN 50 mg QW/QW (N=137)
Injection site erythema (General disorders) | 0 | 1
Injection site pruritus (General disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1
Dengue fever (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Transaminases increased (Investigations) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Demyelinating polyneuropathy (Nervous system disorders) | 1 | 0
Dysaesthesia (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Libido decreased (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ETN 50 mg BW/QW (N=136) | ETN 50 mg QW/QW (N=137)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 1
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 2
Asthenopia (Eye disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 2
Eye discharge (Eye disorders) | 1 | 0
Eye pruritus (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anal inflammation (Gastrointestinal disorders) | 1 | 0
Apical granuloma (Gastrointestinal disorders) | 1 | 0
Chapped lips (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2
Dental caries (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 10
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Gastritis (Gastrointestinal disorders) | 1 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 2 | 0
Lip dry (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 3
Periodontitis (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 1
Cyst (General disorders) | 0 | 1
Fatigue (General disorders) | 8 | 4
Generalised oedema (General disorders) | 1 | 0
Influenza like illness (General disorders) | 2 | 0
Injection site erythema (General disorders) | 7 | 4
Injection site induration (General disorders) | 0 | 1
Injection site oedema (General disorders) | 0 | 1
Injection site pain (General disorders) | 1 | 1
Injection site pruritus (General disorders) | 3 | 0
Injection site reaction (General disorders) | 3 | 7
Injection site swelling (General disorders) | 1 | 2
Malaise (General disorders) | 1 | 2
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 6 | 3
Allergy to arthropod bite (Immune system disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0
Acute tonsillitis (Infections and infestations) | 0 | 1
Body tinea (Infections and infestations) | 0 | 2
Bronchitis (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 3 | 0
Ear infection (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 4 | 0
Fungal infection (Infections and infestations) | 2 | 0
Furuncle (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 2
Infection parasitic (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 2 | 6
Mumps (Infections and infestations) | 1 | 0
Nail infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 14 | 22
Oral herpes (Infections and infestations) | 2 | 1
Otitis externa (Infections and infestations) | 1 | 1
Paronychia (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 6 | 7
Pharyngotonsillitis (Infections and infestations) | 2 | 2
Pneumonia (Infections and infestations) | 1 | 1
Rhinitis (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 1
Tinea cruris (Infections and infestations) | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 9 | 8
Urinary tract infection (Infections and infestations) | 1 | 3
Vaginitis bacterial (Infections and infestations) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 2
Joint sprain (Injury, poisoning and procedural complications) | 2 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 3 | 1
Medical device pain (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase abnormal (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 4
Albumin urine present (Investigations) | 0 | 1
Apolipoprotein B/Apolipoprotein A-1 ratio increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood cholesterol increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 3
Blood insulin increased (Investigations) | 7 | 9
Blood iron decreased (Investigations) | 1 | 0
Blood pressure abnormal (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 0 | 1
Blood triglycerides increased (Investigations) | 2 | 2
C-reactive protein increased (Investigations) | 3 | 0
Glycosylated haemoglobin increased (Investigations) | 1 | 1
Lipids increased (Investigations) | 3 | 3
Liver function test abnormal (Investigations) | 1 | 0
Low density lipoprotein increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0
Prostatic specific antigen increased (Investigations) | 1 | 0
Urine albumin/creatinine ratio increased (Investigations) | 1 | 0
Weight increased (Investigations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 3
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 2 | 0
Myosclerosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 3 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Burning sensation (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0
Dysaesthesia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 15 | 15
Hypersomnia (Nervous system disorders) | 1 | 4
Hypoaesthesia (Nervous system disorders) | 1 | 2
Paraesthesia (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Initial insomnia (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Libido decreased (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Breast pain (Reproductive system and breast disorders) | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 6
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1
Scar pain (Skin and subcutaneous tissue disorders) | 1 | 0
Skin chapped (Skin and subcutaneous tissue disorders) | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0
Skin nodule (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 4
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Wyeth has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.